CLINICAL TRIAL: NCT03265080
Title: A Phase 1 Dose-Escalation Study of ADXS-NEO Expressing Personalized Tumor Antigens, Alone and in Combination With Pembrolizumab in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Study of ADXS-NEO Expressing Personalized Tumor Antigens
Acronym: NEO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Advaxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADXS-NEO-02
Record Dates: First submitted 2017-07-12; First posted 2017-08-29 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Colon Cancer Metastatic; Head and Neck Cancer Metastatic; Metastatic Non-Small Cell Lung Cancer; Urothelial Carcinoma; Metastatic Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Personalized immunotherapy treatment design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): Dose cohorts of 3 participants each will be treated. Initiation of dosing will be staggered by at least 4 weeks for participants in the first cohort, also known as intra-cohort staggering.
  Two dose levels of ADXS-NEO will be explored: 1 x 10^9 and 1 x 10^8 colony forming unit (CFU).
  Interventions: Biological: ADXS-NEO
- Part B (Experimental): Two dose levels of ADXS-NEO will be explored (i.e., 1 x 10^8 and 5 x 10^8 CFU) in combination with 200 mg of pembrolizumab.
  Interventions: Biological: ADXS-NEO; Biological: Pembrolizumab
- Part C (Experimental): ADXS-NEO will be explored at 1 x 10^8 CFU in combination with 200 mg of pembrolizumab in an expansion cohort.
  Interventions: Biological: ADXS-NEO; Biological: Pembrolizumab

INTERVENTIONS:
Biological: ADXS-NEO — Intravenous infusion
Biological: Pembrolizumab — Intravenous infusion
  Arms: Part B; Part C

SUMMARY:
This is a Phase 1, open-label, multicenter study of ADXS-NEO administered alone and in combination with pembrolizumab in participants with select advanced or metastatic solid tumors. This study will be performed in 2 phases, a safety phase (Part A and Part B) and an efficacy phase (Part C).

DETAILED DESCRIPTION:
Mutation-derived tumor antigens, which are often unique to each participant's tumor, represent a new source of targets for cancer immunotherapy. These mutations, which arise during tumorigenesis, are expressed only by the tumor and, as such, may be recognized as newly formed antigens, or neoantigens, by the participant's T cells. The lack of expression of participant-specific tumor mutations in nonmalignant cells suggests that vaccines targeting these tumor mutations have a low risk of autoimmunity and may represent a safer therapeutic approach than many of those currently available. The development of a Listeria monocytogenes (Lm)-based vaccine that expresses these participant-specific tumor antigens and that activates tumor-killing T cells has the potential to be a highly effective form of immunotherapy. In addition, the Lm platform, because it mediates tumor control through multiple mechanisms, may exhibit more robust anti-tumor activity than other vaccine platforms. Thus, the targeting of participant-specific mutation-derived tumor antigens and the concurrent stimulation of host immunity provides a rational approach for boosting anti-tumor immunity, as monotherapy and in combination with anti-programmed cell death protein-1 (PD-1) inhibitors.

ELIGIBILITY:
Inclusion:

1. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
2. Screening tumor biopsy must be adequate for the identification of nonsynonymous somatic mutations (NSMs) by whole exome sequencing and for the development of ADXS-NEO. Biopsies may be repeated for participants whose Screening biopsies are found to be inadequate for the development of ADXS-NEO. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is generally inadequate.
3. Participant population for Part A (ADXS-NEO monotherapy) is as follows:

   1. Histological or cytological diagnosis of metastatic colorectal cancer (CRC) excluding known microsatellite instability (MSI)-high sub-types, metastatic squamous cell carcinoma of head and neck (SCCHN) or metastatic non-small cell lung cancer (NSCLC) that have progressed or have become intolerant to standard therapy, and whose disease may allow management with other available therapies (or a treatment break, if appropriate) for up to approximately 12 weeks following Screening tumor biopsy. More than one form of anti-tumor therapy is allowed during this interval.
   2. For metastatic CRC, up to 4 lines of approved therapy in the advanced or metastatic setting are allowed, including approved antibody and targeted agent therapy. Participants may be eligible if they have received additional lines of therapy upon discussion with and approval by the Sponsor. Participants are excluded if they are known to have MSI-high tumors. If the status of microsatellite stability is not known, participants are eligible. The determination of microsatellite stability for CRC may be made by local testing on any available tissue prior to study entry.
   3. For metastatic SCCHN, up to 2 lines of approved therapy in the advanced or metastatic setting are allowed, including approved antibody therapy and immunotherapy if eligible. Participants may be eligible if they have received additional lines of therapy upon discussion with and approval by the Sponsor.
   4. For metastatic NSCLC, up to 3 lines of approved therapy in the advanced or metastatic setting are allowed, including approved antibodies, targeted agents and immunotherapy if eligible. Tumors harboring squamous and/or non-squamous histologies are eligible. Tumors harboring squamous and/or non-squamous histologies with neuroendocrine or small cell components may be eligible upon discussion with and approval by the Sponsor.
   5. Prior exposure to immunotherapy including, but not limited to, anti-PD1 or anti-Programmed death ligand-1 (PDL-1) antibodies is allowed but not required. Participants who received prior treatment with such agents must meet the following criteria: (a) Full resolution of prior checkpoint inhibitor-related adverse events and no treatment for these adverse events for at least 3 weeks prior to the first infusion of ADXS-NEO; and (b) no history of severe immune related adverse events (irAE) from prior exposure to checkpoint inhibitors. Severe irAEs are defined as any Common Terminology Criteria for Adverse Events (CTCAE) Grade 4 toxicity requiring treatment with corticosteroids or Grade 3 toxicity requiring corticosteroid treatment (greater than 10 mg/day prednisone or equivalent dose) for greater than 12 weeks.
4. Participant population for Part B and Part C (ADXS-NEO + pembrolizumab) is as follows:

   1. Histological or cytological diagnosis of NSCLC, SCCHN, urothelial carcinoma, or melanoma.
   2. Participant has received, and then progressed or been intolerant to up to 3 lines of prior therapy in the advanced or metastatic setting, including approved chemotherapy, targeted therapy, immunotherapy and antibody therapy, if eligible. Participants who have received >3 lines of prior therapy may be eligible upon discussion with and approval by the Sponsor.
   3. For NSCLC: Participants with metastatic NSCLC whose tumors express PD-L1 (tumor proportion score [TPS] ≥1%) as determined by a Food and Drug Administration (FDA)-approved test are eligible, with disease progression on or after platinum-containing chemotherapy. Participants with estimated glomerular filtration rate (EGFR) or anaplastic lymphoma kinase (ALK) genomic tumor aberrations should have disease progression on FDA-approved therapy for these aberrations prior to enrolment.
   4. For SCCHN: participants with recurrent or metastatic SCCHN with disease progression on or after platinum-containing chemotherapy are eligible.
   5. For urothelial carcinoma:

      * Participants with locally advanced or metastatic urothelial carcinoma who are not eligible for cisplatin-containing chemotherapy and whose tumors express PD-L1 [Combined Positive Score (CPS) ≥10] as determined by an FDA-approved test, or participants who are not eligible for any platinum-containing chemotherapy regardless of PD-L1 status, are eligible.
      * Participants with locally advanced or metastatic urothelial carcinoma who have disease progression during or following platinum-containing chemotherapy or within 12 months of neoadjuvant or adjuvant treatment with platinum-containing chemotherapy, are eligible.
   6. For melanoma: participants with unresectable or metastatic melanoma are eligible.
5. Has evaluable or measurable disease for response assessment per RECIST v1.1.
6. Has adequate organ function.
7. Has no major existing comorbidities or medical conditions that will preclude therapy in the view of the Investigator.
8. Baseline blood oxygen saturation on room air of > 95%
9. Resolution to Grade ≤1 by the National Cancer Institute (NCI) CTCAE, Version 4.03 of all clinically significant toxic effects of prior anti-tumor therapy within 3 weeks of first dose of study treatment except for alopecia.
10. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) OR
    2. A WOCBP who agrees to follow the contraceptive guidance during the study treatment period and for at least 120 days after the last dose of study treatment.
11. Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving any dose of ADXS-NEO. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. A male participant is eligible to participate if he agrees to follow the contraceptive guidance during the study treatment period and for at least 120 days after the last dose of study treatment.
13. Provide written informed consent for the trial including mandatory biopsy of accessible lesion(s) during Screening (Parts A, B and C), and mandatory on-treatment biopsy (Parts A and B; if there is no complete resolution of lesions and if the safety risk for biopsy remains acceptable).

Exclusion:

1. Has a newly diagnosed tumor and a curative treatment option or approved therapy is available.
2. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided that they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to first dose of ADXS-NEO (Part A) or pembrolizumab (Part B and Part C). If a participant does not meet these criteria, the participant may be eligible upon discussion and agreement between the Sponsor and Investigator based upon the participant's specific case.
3. Any active autoimmune disease or a documented history of autoimmune disease, or history of a syndrome that required systemic steroids or immunosuppressive medications, except for participants with Grade ≤2 vitiligo or resolved childhood asthma/atopy or uncomplicated dermatitis.
4. History of recently (within previous 12 months) active diverticulitis, symptomatic peptic ulcer disease, colitis, inflammatory bowel disease or any gastrointestinal diseases that, in the opinion of the Investigator and Sponsor's medical monitor would pose a risk to the participant safety.
5. History of other active malignancy for < 2 years prior to enrollment. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cancer that has undergone potentially curative therapy or is felt by the Investigator to be at low risk for recurrence is allowed.
6. History or evidence of cardiovascular risk including any of the following:

   1. History or evidence of clinically significant arrhythmias (ventricular fibrillation, ventricular tachycardia, supraventricular tachycardia, atrial tachycardia/flutter, atrial fibrillation with rapid ventricular response, second or third degree atrioventricular block, and sick sinus syndrome).

      Exception: Participants with controlled atrial fibrillation for >30 days prior to enrollment are eligible. Controlled atrial fibrillation is defined as atrial fibrillation with no ventricular response which requires no change in medication/dosage or addition of new medication or hospital admission within 30 days prior to enrollment.
   2. History of acute coronary syndromes (e.g., myocardial infarction and unstable angina) and/or coronary angioplasty within 6 months prior to enrollment.
   3. History or evidence of Class ≥II congestive heart failure as defined by New York Heart Association (NYHA).
   4. Chronic hypertension (defined as a systolic blood pressure >140 mm Hg and/or diastolic blood pressure >90 mm Hg which cannot be controlled by anti-hypertensive therapy).
   5. Participants with intra-cardiac defibrillators.
   6. Abnormal cardiac valve morphology (Grade ≥2). Participants with grade 1 abnormalities can be entered on study. Participants with moderate valvular thickening should not be entered on study. History of arterial thrombosis (e.g., stroke or transient ischemic attack) in the past 3 months.
7. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
8. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the Screening visit(s) through 120 days after the last dose of study treatment.
9. Active infection requiring systemic therapy or is dependent on or currently receiving antibiotics that cannot be discontinued before dosing. (NOTE: Participants who discontinue an antibiotic prior to dosing must wait at least 5 half-lives after the last dose of antibiotic before receiving ADXS-NEO (Part A) or pembrolizumab (Part B and Part C).
10. Treatment with immune modulators including, but not limited to, chronic immunosuppressive dose of corticosteroid (>10 mg/day of prednisone or equivalent), cyclosporine, or tacrolimus within 4 weeks prior to enrollment. If the participant was receiving corticosteroids, taper or discontinuation must be completed at least 1 week prior to the first dose of ADXS-NEO (Part A) or pembrolizumab (Part B and Part C). Occasional topical corticosteroids and/or inhaled corticosteroids are allowed for a dose equivalency of ≤10 mg prednisone taken orally per week.
11. Known allergy to any component of the study treatment formulation(s).
12. Known history of human immunodeficiency virus (HIV).
13. Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., Hepatitis C virus ribonucleic acid [HCV RNA] [qualitative] is detected).
14. Implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, defibrillators, orthopedic screw[s], metal plate[s], bone graft[s], or other implant[s]). NOTE: More common devices and prosthetics that include arterial and venous stents, dental and breast implants, urinary catheters, and venous access devices (e.g., Port-a-Cath or Mediport) are permitted. The Sponsor must be contacted prior to consenting any participant who has any other device and/or implant.
15. Contraindication (i.e., documented sensitivity/allergy) to trimethoprim/sulfamethoxazole and ampicillin.
16. Contraindication to non-steroidal anti-inflammatory drugs (NSAIDs).
17. In the opinion of the investigator, participant has rapidly progressing disease, OR has life expectancy <6 months, OR would be unable to receive at least one dose of ADXS-NEO.

    Prior/Concomitant Therapy
18. Monoclonal antibody or biologic therapy within 5 half-lives or 28 days, whichever is shorter, prior to first dose of ADXS-NEO (Part A) or pembrolizumab (Part B and Part C). Participants undergoing therapy with pembrolizumab at the time of Screening (Part B) may continue pembrolizumab without the above-mentioned washout period if stable.
19. Received anticancer chemotherapy, surgical treatment, and/or radiation therapy (except palliative radiation therapy for disease-related pain in consultation with the Sponsor's medical monitor) within 3 weeks of first dose of ADXS-NEO (Part A) or pembrolizumab (Part B and Part C).
20. Because of a possible interaction between attenuated Lm and phosphoinositide 3-kinases (PI3K) inhibitor (may be directly involved in regulation of TNFα production and enhance Lm virulence), participants receiving a PI3K or TNFα inhibitor within 3 weeks of first dose of study treatment, or are expected to receive such agents at any time during the treatment period, are excluded.
21. Received a live vaccine within 30 days prior to the first dose of ADXS-NEO (Part A) or pembrolizumab (Part B and Part C).
22. Major surgery, including surgery for a new artificial implant and/or medical device, which is permitted by the protocol, within 6 weeks prior to initiation of ADXS-NEO (Part A) or pembrolizumab (Part B and Part C). NOTE: All toxicities and/or complications must have recovered to baseline or Grade 1 prior to the initiation of study treatment. Consult with the Sponsor prior to enrolling participants who recently had major surgery or who have a new artificial implant, and/or devices.

    Prior/Concurrent Clinical Study Experience
23. Currently participating in or has participated in a study of an investigational agent or is using an investigational device within 3 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From the first dose up to 20 months
Maximum tolerated dose | 4 weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline to measured progressive disease or start of new anticancer therapy (approximately 15 months)
ORR According to immune Response Evaluation Criteria in Solid Tumors (iRECIST) | Baseline to measured progressive disease or start of new anticancer therapy (approximately 15 months)
Disease Control Rate (DCR) According to RECIST v1.1 | Baseline to measured progressive disease or death due to any cause (approximately 15 months)
DCR According to iRECIST | Baseline to measured progressive disease or death due to any cause (approximately 15 months)
Duration of Response (DoR) According to RECIST v1.1 | Baseline to measured progressive disease or death due to any cause (approximately 15 months)
DOR According to iRECIST | Baseline to measured progressive disease or death due to any cause (approximately 15 months)
Progression Free Survival (PFS) According to RECIST v1.1 | Baseline to measured progressive disease or death due to any cause (approximately 15 months)
PFS According to iRECIST | Baseline to measured progressive disease or death due to any cause (approximately 15 months)
Overall Survival | Baseline to death due to any cause (approximately 20 months)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Honor Health, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - Ochsner Clinic Foundation - Ochsner Cancer Institute, New Orleans, Louisiana
  - Atlantic Health System, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hecht JR, Sheeri S, Heyburn J, Parsi M , Gutierrez AA, Tsai F. Clinical and immunogenicity data of a personalized neoantigen-Listeria vaccine in cancer patients: preliminary results. IO Combinations 360. Philadelphia, PA 20 June 2019.
- [Result] Tsai F, Goldman JW, Kosoff R, Heyburn JW, Sands T, Sheeri S, Petit R, Gutierrez AA, Hecht JR. Safety and Immunogenicity of a Personalized Neoantigen-Listeria Vaccine in Cancer Patients. Frontiers in Cancer Immunotherapy, The New York Academy of Sciences, May 14-15, 2019,New York, NY
- [Result] Hecht JR, Goldman JW, Hayes S, Balli D, Princiotta MF, Dennie JG, Heyburn J, Sands T, Sheeri S, Petit R, Gutierrez AA, Tsai F. Safety and immunogenicity of a personalized neoantigen -Listeria vaccine in cancer patients. AACR Annual Meeting 2019.